CLINICAL TRIAL: NCT06016400
Title: A Randomized, Double-blind, Single-center Clinical Trial of Using Vitamin D to Reduce Oral Mucosal Inflammation in Chemotherapy Patients With Oral Squamous Cell Carcinoma
Brief Title: Using Vitamin D to Reduce Oral Mucosal Inflammation in Chemotherapy Patients With Oral Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-KY-049
Record Dates: First submitted 2023-08-07; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Oral Squamous Cell Carcinoma; Oral Mucositis
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Stomatitis | interventions — alfacalcidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Alfacalcidol Drops,1ug a day,40day
  Interventions: Drug: Alfacalcidol Oral Solution
- control group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alfacalcidol Oral Solution — Alfacalcidol Oral Solution 1ug a day
  Arms: intervention group
Drug: Placebo — Placebo
  Arms: control group

SUMMARY:
Oral squamous cell carcinoma is the most common malignant tumor of the oral and maxillofacial region. Currently, surgery is the main method of comprehensive treatment. TPF (paclitaxel, cisplatin, and fluorouracil) chemotherapy regimen is one of the important methods for the treatment of oral squamous cell carcinoma. Adjuvant chemotherapy before and after surgery can significantly improve the therapeutic effect of oral cancer patients. Oral mucositis (OM) is a common side effect during chemotherapy, which seriously affects the quality of life of chemotherapy patients and may lead to the termination of chemotherapy. Prevention and treatment of oral mucositis is still an urgent clinical problem. Investigators' previous studies have found that vitamin D can significantly inhibit the proliferation, migration, invasion and metastasis of oral squamous cell carcinoma cells, and vitamin D can protect normal oral mucosal tissue by inhibiting pyroptosis caused by platinum-based chemotherapy drugs. Based on the previous basic research, this project intends to conduct a single-center, prospective, clinical randomized controlled study on the clinical efficacy of vitamin D in reducing oral mucosal inflammation in patients with oral squamous cell carcinoma undergoing TPF chemotherapy, in order to provide evidence-based medical evidence for the clinical use of vitamin D in reducing oral mucosal inflammation in patients with oral cancer chemotherapy. The results of this study are expected to serve as guidelines to guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20-70 years
2. Patients with pathologically diagnosed oral squamous cell carcinoma who need TPF-based chemotherapy regimens, and whose expected survival time is greater than 6 months
3. Patients whose serum 25-hydroxyvitamin D level was vitamin D deficiency (<30nmol/L) and adequate (30-50nmol/L) before chemotherapy
4. Patients and their families agree to participate in this trial and sign an informed consent form
5. No cognitive impairment

Exclusion Criteria:

1. People with oral ulcers or other oral mucosal diseases (such as: oral mucosal pemphigus, etc.) at the beginning of the study
2. Patients who are allergic to alfacalcidol drops
3. Patients with severe cardiac insufficiency, liver and kidney insufficiency, and systemic infectious diseases
4. Pregnant women (judged by HCG test) and lactating patients
5. Participating in other clinical trials during the study
6. Those who do not understand or cooperate with clinical trials
7. Patients with hypervitaminosis D, hypercalcemia, hyperphosphatemia and renal rickets

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Within two months from the start of chemotherapy | Within two months from the start of chemotherapy
  Oral mucosal hyperemia, erythema, erosion, ulceration and fibrosis appear, accompanied by clinical manifestations such as pain, difficulty eating, dry mouth, and taste disturbance.

SECONDARY OUTCOMES:
Grading of oral mucositis in patients treated with vitamin D and placebo | Within two months from the start of chemotherapy
  According to the American Oncology Nurse Oral Mucositis Evaluation Scale, the score <8 is normal; 9-10 is mild; 11-12 is moderate; >12 is severe
Changes in the quality of life of patients in vitamin D treatment group and placebo group before | Within two months from the start of chemotherapy
  University of Washington quality of life scale
Healing time of oral mucositis in vitamin D treatment group and placebo group | Within two months from the end of chemotherapy
  Time to cure of patients with oral mucositis
Length of hospital stay of patients in vitamin D treatment group and placebo group | Within two months from the start of chemotherapy
  Length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No